CLINICAL TRIAL: NCT04858724
Title: Construction of a Multi-center Database for Primary IgA Nephropathy
Brief Title: The Chinese Registry of Prognostic Study of IgA Nephropathy (CRPIGA)
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Collaborators: RenJi Hospital (Other); Huashan Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: CRPIGA
Record Dates: First submitted 2021-04-19; First posted 2021-04-26 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: IgA Nephropathy
Keywords: IgAN; database; multicenter
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Establish an IgAN cohort collaboration group and expert committee to carry out registration research.
2. Construct IgAN structured data set standards, formulate structured data collection templates of diagnosis and treatment , and establish multi-center data integration systems on this basis.
3. Establish a standardized IgAN database for combined Hospital Information System and the big data platform of the Medical Federation.
4. Develop IgAN database managements and open standards for data sharing, and carry out high-quality clinical or basic research.

DETAILED DESCRIPTION:
Primary IgA nephropathy (IgAN) is the most common form of glomerulonephritis in China and the world. It is the main reason for Chinese young people's renal failure. The main difficulties in clinical IgAN and treatment are 1) high clinical and prognostic heterogeneity, the prognosis cannot be accurately predicted; 2) no clinically available biomarkers, diagnosis is established by kidney biopsy; 3) The lack of specific treatment methods. These lead 20-40% of IgAN patients to develop end-stage renal failure (ESRD) after 10 to 20 years. Therefore, to improve clinical diagnosis, treatment, and scientific research of IgAN, it is much-needed to establish high-quality long-term cohort study, multi-center database, biobank, and conduct high-quality clinical research.

The incidence of IgAN in the Asia Pacific region is higher than in other regions, and China is one of the countries with the highest incidence of IgAN in the world. Although the number of IgAN patients in our country is vast and the clinical data and patient sample resources are abundant, the clinical diagnosis and treatment are not standardized, the follow-up rate is low, and the quality of clinical data is poor, which seriously affect the development of related clinical research. Therefore, optimization and integration of health care big data under careful top-level design is urgently needed.

Regarding IgAN, the Nephrology Department of Ruijin Hospital has been active in clinical database construction and clinical biobank management and has carried out several clinical and basic research. The world's largest IgAN cohort-CRPIGA cohort has been established, all patients in the cohort are followed up in a standardized manner by special personnel, and the data is recorded in a clinical database in real-time. However, optimization and integration of health care big data under careful top-level design is urgently needed. It is to establish IgAN specific disease structured data set standard in a multi-center linkage mode, formulate IgAN diagnosis and treatment specifications and clinical pathway standards, develop structured clinical case diagnosis and treatment information collection template, real-time scrape the actual clinical IgAN diagnosis and treatment data of various hospitals through the big data platform of health care consortium, clean and structure the acquired data, establish a multi-center structured database, integrate resources, strengthen advantages, and provide a qualified database for clinical research in the real world. All diagnosis and treatment data for the same patient are linked and integrated to offer individual patient-based longitudinal tracking records and support evidence-based medicine.

This study aims to improve the scale and quality of the IgAN multi-center cohort database, advance the clinical and basic research of IgAN, standardize and optimize the clinical diagnosis and treatment path of IgAN, provide more effective and safe treatment options for more IgAN patients and also provide evidence-based medicine evidence support.

ELIGIBILITY:
Inclusion Criteria:

1. No age limit, no gender limit;
2. Kidney biopsy confirmed primary IgA nephropathy;
3. Sign the informed consent form voluntarily

Exclusion Criteria:

1. IgA nephropathy is secondary to systemic diseases such as systemic lupus erythematosus and allergic purpura;
2. IgAN is clinically diagnosed but not confirmed by pathology;
3. The patient refuses to participate;
4. Patients judged by other investigators to be unsuitable for inclusion in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Biopsy-proven primary IgAN patients
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of a decline in estimated glomerular filtration rate by > 50% from baseline | 1 year
  To evaluate the renal function
The proportion of doubling serum creatinine compared with baseline | 1 year
  To evaluate the renal function
Incidence of ESRD | 1 year
  To evaluate the renal function

SECONDARY OUTCOMES:
Incidence of cardiovascular events | 1 year
  Record of Cardiovascular events during follow-up period
Incidence of All-cause death | 1 year
  Record of All-cause death during follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Xie, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China